CLINICAL TRIAL: NCT05040425
Title: Radioprotective Effect of Chinese Herbal Medicine on Ionizing Radiation-Induced Oral Mucositis
Brief Title: Radioprotective Effect of Chinese Herbal Medicine on Oral Mucositis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Research Institute of Chinese Medicine, Ministry of Health and Welfare (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202101231A3
Record Dates: First submitted 2021-09-03; First posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-08

CONDITIONS: Head and Neck Cancer; Oral Mucositis
Keywords: Oral mucositis; Radiotherapy; Head and neck cancer; Chinese herbal medicine; Randomized trial
MeSH Terms: conditions — Head and Neck Neoplasms; Stomatitis

STUDY DESIGN:
Intervention Model Description: The participants selected at screening who provide written informed consent will be randomly allocated to two groups. One will be submitted to Chinese herbal medicine group, and the other to control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chinese herbal medicine treatment (Experimental)
  Interventions: Drug: Zi-Yin-Liang-Ge-San
- Non-Chinese herbal medicine treatment (No Intervention)

INTERVENTIONS:
Drug: Zi-Yin-Liang-Ge-San — Zi-Yin-Liang-Ge-San is composed of five herb ingredients, namely Rx. Scutellariae (Huang Qin), Rx. Glycyrrhizae (Gan Cao), Hb. Dendrobii (Shi Hu), Rx. Ophiopogonis (Mai Men Dong), and Hb. Menthae Haplocalycis (Bo He). It is orally administrated trice daily from the first day to the end of RT in the treatment group, aiming to prevent and manage the OM. ZYLGS is manufactured as a concentrated herbal extract, constituted 4 g per packet, and origin from pharmaceutical companies in Taiwan with good manufacturing practice (GMP).
  Arms: Chinese herbal medicine treatment

SUMMARY:
This protocol describes a randomized, double-arm, parallel-group, open-label controlled study that aims to evaluate the efficacy of Chinese herbal medicine on head and neck cancer patients with oral mucositis toxicities and quality of life during radiotherapy.

DETAILED DESCRIPTION:
200 head and neck cancer patients who were scheduled for radiotherapy are randomly assigned at a 1:1 ratio to two arms: control group and those treated with Zi-Yin-Liang-Ge-San containing Rx. Scutellariae, Rx. Glycyrrhizae, Hb. Dendrobii, Rx. Ophiopogonis, and Hb. Menthae Haplocalycis from day 1 of radiotherapy. The study lasted at least 6 weeks and the clinical benefit was determined by onset, gradation of mucositis (Common Terminology Criteria for Adverse Events v5.0), oral pain (visual analysis scale) for each week during RT. Nutritional status, EORTC Quality of Life Core Questionnaire (QLQ-C30) and head and neck module (QLQ-H&N35), Body Constitution Questionnaire (BCQ), and electrical body conductivity were evaluated before and after radiotherapy. Patient-Reported Outcomes version of Common Terminology Criteria for Adverse Events (PRO-CTCAE), serious adverse events, blood and biochemical analysis will be recorded to evaluate the safety.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven stage II-IV squamous HNC
* Indication for radiotherapy or radio-chemotherapy
* No history of antitumor therapies
* No history of oral ulcer and salivary gland diseases
* Normal vital signs (body temperature: 36 to 37.5∘C, heart rate: 60 to 100 beats per minute, respiratory rate: <20 per minute, and mean arterial pressure: 70 to 100mmHg), and Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2

Exclusion Criteria:

* Terminal cancer for which aggressive treatments were not suitable
* Impaired renal or hepatic function at initial diagnosis (including chronic kidney disease stages III, IV, and V and Aspartate transaminase (AST), Alanine aminotransferase (ALT) ≥5 × the upper normal limit)
* Uncontrolled psychiatric problems or altered mental status
* Had received medications for other clinical trials

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-08-30 (Estimated); Primary Completion 2022-08-17 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Degree of oral mucositis | During the radiotherapy course, up to 6 weeks
  The degree was graded by the NHI Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0)
Mucositis pain | During the radiotherapy course, up to 6 weeks
  100-mm-visual analog scale (VAS, 0-100)

SECONDARY OUTCOMES:
Health related-QoL (1) | Baseline, 4th week, and 6th week of radiotherapy completion
  EORTC Core Quality of Life questionnaire (EORTC QLQ-C30)
Health related-QoL (2) | Baseline, 4th week, and 6th week of radiotherapy completion
  Quality of Life Head and Neck Module (QLQ-H&N35)
Body mass index (BMI) | During the radiotherapy course, up to 6 weeks
  Body mass index (BMI)

OTHER OUTCOMES:
Traditional Chinese medicine constitution | Baseline, 4th week, and 6th week of radiotherapy completion
  Body Constitution Questionnaire (BCQ)
Electrical body conductivity | Baseline, 4th week, and 6th week of radiotherapy completion
  Meridian Energy Analysis Device

IPD SHARING:
Plan to Share IPD: No
The datasets during and/or analyzed during the current study available from the corresponding author on reasonable request.